CLINICAL TRIAL: NCT04140578
Title: Antibiotic Prophylaxis in Patients Undergoing Endoscopic Injection of Cyanoacrylate for Primary and Secondary Prevention of Gastric Variceal Bleeding
Brief Title: Antibiotic Prophylaxis in Patients Undergoing GVO
Acronym: ABX-GV
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2017-01-027C
Record Dates: First submitted 2019-08-29; First posted 2019-10-28 (Actual); Last update posted 2019-10-28 (Actual); Status verified 2019-10

CONDITIONS: Gastric Varix; Sepsis; Liver Cirrhoses; Fever
Keywords: Gastric variceal rebleeding; Sepsis; cyanoacrylate injection
MeSH Terms: conditions — Esophageal and Gastric Varices; Sepsis; Fever | interventions — Ertapenem

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Antibiotic (Experimental): Participate will be acepted ertapenem(1g) iv before endoscopic cyanoacrylate injection obliteration
  Interventions: Drug: Ertapenem
- Control (No Intervention): Participate will not be acepted ertapenem(1g) iv before endoscopic cyanoacrylate injection obliteration

INTERVENTIONS:
Drug: Ertapenem — inject from iv drip before endoscopic cyanoacrylateinjection obliteration
  Other Names: Invanz
  Arms: Antibiotic

SUMMARY:
We design a randomized trial to clarify the necessity of antibiotic prophylaxis for the patients chronic liver disease with gastric varices treated by elective GVO.

DETAILED DESCRIPTION:
Gastric varices is not uncommon is patients with chronic liver diseases including liver cirrhosis and hepatocellular carcinoma. Occurrence of gastric varices (GV) rupture is less often than esophageal varices (EV) but it is characteristic of higher rebleeding rate and mortality and represents an even tougher problem than EV hemorrhage. Endoscopic treatment is an alternative in the management of GV bleeding. Injection sclerotherapy has been applied to arrest GV hemorrhage but it is associated with a high rebleeding rate (50~90%) and thus is regarded as only a temporary hemostatic measure. The advantage of endoscopic variceal ligation is not suggested due to its high rebleeding rate more than 50%. Endoscopic injection of N-butyl-2-cyanoacrylate, a so-called "tissue glue",is more effective to treat GV bleeding because of more than 90% successful rate to arrest acute bleeding. The theoretical advantages of tissue glue derives from its unique ability to plug the varix lumen immediately after injection into varices. However, its rebleeding rate is still high around 30~40% and has potential treatment-related morbidity such as embolic and septic complications. Regardless of these disadvantage, the guideline form major international society and Bavenoconsensus recommend GVO as the first treatment of choice for GV bleeding. Therefore how to prevent the potential complications and reduce rebleedingremains an important and practical issue.

With regarding to potential septic infections and rebleeding, the effects of impaired leukocyte function in cirrhotic patients and reduced immunity and increased gut permeability of severe hemorrhagic patients were contributory. In these immunocompromised hosts, when invasive procedure such as GVO is deployed for these patients, the septic complication become un-neglectable, We found (Gastrointest Endosc 2001) more than 1/3 patients undergoing GVO may complicated with bacteremia. Although most of these bacteremia were self-limited, 2% died of sepsis. Moreover, lots of cases were reported due to persistent and recurrent bacterial infections caused by GVO. Antibiotic prophylaxis has been suggested as an integral part for the management of cirrhotic patients with acute varicealbleeding by major international society and Baveno consensus. However, there is no evidence to suggest antibiotic prophylaxis for the patients treated by elective GVO. Therefore we design a randomized trial to clarify the necessity of antibiotic prophylaxis for the patients chronic liver disease with gastric varices treated by elective GVO.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with live cirrhosis and/or hepatoma
2. Aged 20 to 85, who had endoscopy-treatment EV(-)GV(+)or EV<GV

Exclusion Criteria:

1. Had a terminal illness of any major organ system,such as heart failure, kindey failure,COPD
2. Patients recieve antibiotics recently.
3. Patients suspected infection.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2017-01-28 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevetion of sepsis | 3 years
  If Antibiotic Prophylaxis can reduce sepsis in Patients Undergoing GVO

SECONDARY OUTCOMES:
Rebleeding rate | 3 years
  If Antibiotic Prophylaxis can reduce GV rebleeding rate
Pevention of Refractory bacterial infection | 3 years
  If Antibiotic Prophylaxis can reduce infection rate in Patients Undergoing GVO
Mortality | 3 years
  If Antibiotic Prophylaxis can decrease mortality in Patients Undergoing GVO

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Chih Hou, Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Veteran General Hospital-Taipei, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No